CLINICAL TRIAL: NCT05820308
Title: Feasibility and Acceptability of a Randomized Controlled Trial Comparing a Companion Dog-Walking Intervention to an Attention Control Education Intervention on the Psychological Health of Adult Intensive Care Unit Survivors
Brief Title: Companion Dog Walking for ICU Survivor Health
Acronym: POOCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri, Kansas City (Other)
Collaborators: Sigma Theta Tau International Honor Society of Nursing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2094468
Record Dates: First submitted 2023-03-28; First posted 2023-04-19 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Post Intensive Care Syndrome; Depression; Anxiety; Quality of Life
Keywords: Post Intensive Care Syndrome; ICU Survivors; Companion dog; Depression; Anxiety; Quality of life
MeSH Terms: conditions — postintensive care syndrome; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be randomly assigned and masked to their group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Companion dog walking
  Interventions: Behavioral: Companion Dog Walking
- Attention Control Group (Active Comparator): Educational resources about dog health
  Interventions: Behavioral: Attention Control Group

INTERVENTIONS:
Behavioral: Companion Dog Walking — Participants will be asked to walk their dog three times per week, for a minimum of 30 minutes each day of walking, over an 8-week period.
  Arms: Intervention Group
Behavioral: Attention Control Group — Participants will be asked to read educational materials on dog health once per week, over an 8-week period.
  Arms: Attention Control Group

SUMMARY:
The goal of this clinical trial is to determine the feasibility and acceptability of a randomized controlled trial comparing a pet dog walking intervention to an attention control education intervention in adult intensive care unit survivors.

The main question[s] it aims to answer are:

* What is the feasibility of a pet dog-walking intervention compared to an attention control education intervention on depression, anxiety, cortisol, and quality of life for adult ICU survivors.
* What is the acceptability of a pet dog-walking intervention compared to an attention control education intervention on depression, anxiety, cortisol, and quality of life for adult ICU survivors.

The secondary question[s] it aims to answer are:

- What are the differences in depression, anxiety, serum cortisol, and quality of life between and within a companion dog walking intervention compared to an attention control education intervention for ICU survivors?

Participants in the intervention group will be asked to:

* Participate in dog walking with their pet dog at least three times per week, for at least 10 minutes each walk, for 8-weeks.
* Wear an activity monitor and record their dog walks in a diary.
* Complete surveys to measure depression, anxiety, and quality of life at the start of the study, after week 4, and after week 8.
* Have blood drawn to measure cortisol levels at the start of the study, after week 4, and after week 8.

Participants in the control group will be asked to:

* Read educational materials about their pet dog's health once every week (education materials are provided by the researchers).
* Wear an activity monitor and record when they read their education materials in a diary.
* Complete surveys to measure depression, anxiety, and quality of life at the start of the study, after week 4, and after week 8.
* Have blood drawn to measure cortisol levels at the start of the study, after week 4, and after week 8.

Participants will be assigned to an intervention group or a control group to see if there are differences in depression, anxiety, serum cortisol, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years)
* ICU survivors (spent ≥24 hours in the ICU)
* Will be discharged directly home from hospital.
* Able to speak, read, and understand English
* Physically capable of dog walking
* Individuals who have symptoms of depression and/or anxiety
* Individuals who own a companion dog and walk their dog <10 minutes/week
* Participants scoring ≤ 20 seconds on the TUG Test

Exclusion Criteria:

* Individuals at high risk for suicide
* Individuals with severe depression or anxiety
* Individuals who recently started treatment for depression and/or anxiety
* Individuals with cognitive impairment
* Dog walking is deemed unsafe with and for the dog
* Medical Provider authorization is indicated but not provided
* Individuals who live outside a 45-mile radius of Colorado Springs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Study Feasibility as assessed by recruitment results, attrition rates, intervention fidelity, and missing data points | Feasibility data will be collected and analyzed from the time identifying, screening, and recruiting eligible participants begins to the time the final participant completes the study; no more than 12 months.
  Data will be collected to answer the following questions:
  1. To what extent does the recruitment procedure produce study participants?
  2. How many participants met inclusion and exclusion criteria?
  3. What are the obstacles to recruitment?
  4. What was the attrition rate of participants?
  5. To what extent was fidelity of the intervention maintained by participants?
  6. To what extent were measurements completed?
  7. What was the extent and patterns of missing data?
Study Acceptability as assessed by participant responses to survey questions regarding the amount of time spent in the study, the measurement tools used, the masking procedure, and the intervention. | Acceptability will be assessed post-intervention after participants complete the 8-week study period.
  Participants will complete an exit survey and will be asked to report on: (1) the acceptability of the time spent in the study and per session, (2) the acceptability of completing the measurement tools, (3) the acceptability of the masking procedure, (4) the acceptability of the intervention, (5) if they intend to continue the intervention after the end of the study, and (6) to report any suggestions for improvement they have.

SECONDARY OUTCOMES:
Change in Depression | Depression will be measured at baseline, half way through the intervention (at the end of week 4), and post intervention (at the end of week 8).
  The Center for Epidemiologic Studies Depression Scale is a 20-item self-report tool that assesses intensity of depression using a 4-point Likert scale. Lower scores indicate milder levels of depression while higher scores indicate more severe depression (potential score 0-60). Clinically meaningful depression is represented by a score of 16 or greater.
Change in Anxiety | Anxiety will be measured at baseline, half way through the intervention (at the end of week 4), and post intervention (at the end of week 8).
  The Spielberger State Trait Anxiety Inventory is a 40-item self-report assessment tool using a 4-point Likert scale that assesses both trait and state anxiety. The higher a participant's score (potential score 20-80 on each subscale) the higher the level of anxiety. No/low anxiety = 20-37 points; moderate anxiety= 38-44 points; and high anxiety=45-80 points, with a cut-off point of 39 indicting clinically significant symptoms of anxiety.
Change in Quality of Life as assessed by health related quality of life indicators including physical functioning, physical and emotional limitations, social functioning, bodily pain, general and mental health. | Quality of life will be measured at baseline, half way through the intervention (at the end of week 4), and post intervention (at the end of week 8).
  The Short Form 36 is a 36-item self-report questionnaire using various ranking questions to measure health related quality of life. The Shot Form 36 examines eight dimensions of health related quality of life (physical functioning, physical and emotional limitations, social functioning, bodily pain, general and mental health). The higher the score (max score =100) the better the health and wellbeing, the lower the score (minimum score=0) the poorer the health and wellbeing.
Change in Serum Cortisol | Serum Cortisol will be measured at baseline, half way through the intervention (at the end of week 4), and post intervention (at the end of week 8).
  Peripheral venous blood samples will be obtained from participants or analysis at a laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Nelson, MSN, RN, Principal Investigator — University of Missouri, Kansas City
Locations (2):
- United States (2):
  - Penrose Hospital, Colorado Springs, Colorado
  - St. Francis Hospital, Colorado Springs, Colorado

IPD SHARING:
Plan to Share IPD: No